CLINICAL TRIAL: NCT01917708
Title: Abatacept for Post-Transplant Immune Suppression in Children and Adolescents Receiving Allogeneic Hematopoietic Stem Cell Transplants for Non-Malignant Diseases
Brief Title: Bone Marrow Transplant With Abatacept for Non-Malignant Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Horan, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00069836
Record Dates: First submitted 2013-07-24; First posted 2013-08-07 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Hurler Syndrome; Fanconi Anemia; Glanzmann Thrombasthenia; Wiskott-Aldrich Syndrome; Chronic Granulomatous Disease; Severe Congenital Neutropenia; Leukocyte Adhesion Deficiency; Shwachman-Diamond Syndrome; Diamond-Blackfan Anemia; Dyskeratosis-congenita; Chediak-Higashi Syndrome; Severe Aplastic Anemia; Thalassemia Major; Hemophagocytic Lymphohistiocytosis; Sickle Cell Disease
Keywords: non malignant conditions; blood and marrow transplant
MeSH Terms: conditions — Mucopolysaccharidosis I; Fanconi Anemia; Thrombasthenia; Wiskott-Aldrich Syndrome; Granulomatous Disease, Chronic; Neutropenia, Severe Congenital, Autosomal Recessive 3; Leukocyte adhesion deficiency type 1; Shwachman-Diamond Syndrome; Anemia, Diamond-Blackfan; Dyskeratosis Congenita; Chediak-Higashi Syndrome; Anemia, Aplastic; beta-Thalassemia; Lymphohistiocytosis, Hemophagocytic; Anemia, Sickle Cell | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abatacept (Experimental): 4 doses of abatacept 10 mg/kg/dose will be given on days -1, +5, +14, and +28.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — All patients will receive 4 doses of abatacept in addition to standard GVHD prophylaxis with cyclosporine and mycophenolate mofetil.
  Other Names: Orencia

SUMMARY:
This is a single arm, phase I study to assess the tolerability of abatacept when combined with cyclosporine and mycophenolate mofetil as graft versus host disease prophylaxis in children undergoing unrelated hematopoietic stem cell transplant for serious non-malignant diseases as well as to assess the immunological effects of abatacept. Participants will be followed for 2 years.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) represents the only viable cure for children who suffer from a wide variety of rare, serious non-malignant diseases, such as Fanconi Anemia, Hurler syndrome, and hemophagocytic lymphohistiocytosis. A major obstacle to the success of HSCT is morbidity and mortality from graft versus host disease (GVHD), driven by donor T cells recognizing and reacting against disparate host antigens. This trial is being conducted as a step toward testing the long-term hypothesis that the costimulation blockade agent abatacept can be added to a standard post-transplant GVHD prophylaxis regimen, cyclosporine and mycophenolate mofetil, to improve disease-free survival after unrelated hematopoietic stem cell transplantation (HSCT) using reduced intensity conditioning for children with non-malignant diseases (NMD). This study will have the following Specific Aims:

Specific Aim #1: To conduct a multicenter pilot assessing the tolerability of abatacept (n=10). Patients will receive four doses (10 mg/kg IV on days -1, +5, +14 and +28), a schedule well tolerated by adolescents and adults with hematologic malignancies in a previous pilot. Abatacept will be combined with cyclosporine and mycophenolate mofetil.

Specific Aim #2: To examine the immunological effects of abatacept in this setting.

Three reduced intensity conditioning regimens that have been shown to be effective in achieving sustained engraftment in patients with non-malignant diseases are available for use, depending on the patient's disease:

* Patients with Fanconi anemia will receive fludarabine, low dose cyclophosphamide, and anti-thymocyte globulin.
* Patients with severe aplastic anemia will receive low dose total body irradiation, fludarabine, cyclophosphamide, and anti-thymocyte globulin.
* Patients with other NMD will receive either the low dose total body irradiation regimen or an alemtuzumab, fludarabine, thiotepa, and melphalan regimen.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 0-21 years at the time of admission for transplant.
* Must have one of the following diseases:

  1. Glanzmann thrombasthenia
  2. Wiskott-Aldrich syndrome or other combined immune deficiency
  3. Chronic-granulomatous disease
  4. Severe congenital neutropenia (with resistance to granulocyte-colony stimulating factor (GCSF) or chronic requirement of GCSF doses ≥10 mcg/kg)
  5. Leukocyte adhesion deficiency
  6. Shwachman-Diamond syndrome
  7. Diamond-Blackfan anemia ((transfusion dependent, including steroid failure or inability to wean steroids)
  8. Thalassemia major
  9. Fanconi anemia
  10. Hemophagocytic lymphohistiocytosis (inherited or acquired refractory to therapy or with recurrent episodes of hyperinflammation)
  11. Dyskeratosis-congenita
  12. Hurler Syndrome
  13. Chediak-Higashi syndrome
  14. Acquired (immune; non-inherited, non-congenital) severe aplastic anemia
  15. Sickle cell disease (SCD) (Hgb SS or S-Beta 0 thalassemia) will be eligible between ages 3 and 9.99 and with severe disease.
  16. Other inherited or congenital marrow failure syndromes complicated by severe aplastic anemia
  17. Other inherited or congenital red blood cell disorders requiring monthly chronic transfusion therapy.
  18. Congenital platelet disorders requiring frequent platelet transfusions (patient must have received at least 10 transfusions in the last 3 years).
  19. Other inherited or congenital granulocyte disorders resulting in at least three inpatient hospitalizations in the past three years for infection.
* Must have an unrelated adult donor (marrow or PBSC) who is at least a 7/8 match (A, B, C, DRB1; the mismatch can be at an allele or antigen level) or an unrelated cord blood unit that is matched at least seven of eight loci (A, B and C antigen level-DRB1 allele level) and provides a minimum pre-cryopreservation total nucleated cell (TNC) dose of 7.5 x 107 TNC/kg recipient weight. Mismatches at the DRB1 locus may be at an antigen or allele level.

Exclusion Criteria:

* Human leukocyte antigen (HLA) matched related donor.
* Severe combined immune deficiency.
* Bridging (portal to portal) fibrosis or cirrhosis of the liver.
* Pulmonary: diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin), forced expiratory volume (FEV1) or forced vital capacity (FVC) < 40% of predicted. In child unable to perform pulmonary function testing, a chronic need for supplemental oxygen will serve as the exclusionary criterion.
* Severe renal dysfunction defined as estimated glomerular filtration rate (GFR) of <60 ml/min/1.73m2.
* Severe cardiac dysfunction defined as shortening fraction < 25%.
* Neurologic impairment other than hemiplegia, defined as full-scale intelligence quotient (IQ) less than or equal to 70, quadriplegia or paraplegia, inability to ambulate, or any impairment resulting in decline of Lansky performance score to < 70%.
* Clinical stroke within 6 months of anticipated transplant.
* Karnofsky or Lansky functional performance score < 50%
* HIV infection.
* Uncontrolled viral, bacterial, fungal or protozoal infection at the time of study enrollment.
* Patient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate bone marrow transplantation.
* Patient or patient's guardian(s) unable to understand the nature and risks inherent in the blood and marrow transplant process.
* History of non-compliance severe enough in the estimation of the treating team to preclude the patient from undergoing unrelated donor transplantation.
* Patient is pregnant or lactating
* Patients HLA antibody testing demonstrates an antibody directed against a disparate HLA molecule.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Tolerability of Abatacept | 1 year post-transplant
  The primary endpoint for this trial will be tolerability, defined in terms of the success in administering all prescribed doses of abatacept.
  Abatacept will be deemed to be poorly tolerated if any of the following conditions are met:
  * More than one dose is withheld.
  * Death from an infection that occurs within 30 days of receiving the last prescribed dose of abatacept, but that is not preceded by systemic immunosuppressive therapy for GVHD
  * Post-transplant lymphoproliferative disorder (PTLD) that occurs within 100 days of receiving the last prescribed dose, but that is not preceded by systemic immunosuppressive therapy for GVHD.
  If less than 4 patients (of at least 18 evaluable patients) tolerate abatacept poorly, abatacept will be deemed tolerable. If there are fewer than 18 evaluable patients, if 3 of the first 10 patients treated tolerate abatacept poorly, abatacept will be deemed tolerable.

SECONDARY OUTCOMES:
Proportion of Participants Experiencing Regimen-related Toxicity (RRT) | Day 42 post-transplant
  Regimen-related toxicity is scored according to the Bearman scale. Major RRT, defined as grade 4 (causing death) in any organ system or grade 3 for pulmonary, cardiac, renal, oral mucosal, neurologic or hepatic, will be recorded.
Days until Neutrophil Recovery | 1 year post-transplant
  Neutrophil recovery is defined as the first of 3 consecutive days following the nadir that the absolute neutrophil count is at least 500/µl.
Days until Platelet Recovery | 1 year post-transplant
  Platelet recovery is defined as the first day that the platelet count is at least 20 thousand/µl without a transfusion in the preceding 7 days.
Number of Participants with Non-engraftment | 1 year post-transplant
  Non-engraftment is defined as lack of neutrophil recovery (defined as absolute neutrophil count (ANC )>0.5 *109/L for three consecutive days) by 28 days post-transplant or neutrophil recovery with lack of myeloid donor chimerism.
Number of Participants with Secondary Graft Failure | 1 year post-transplant
  Secondary graft failure is defined by initial engraftment but subsequent development of an ANC <0.5*109/L for fourteen consecutive days.
Number of Participants with Graft Loss | 1 year post-transplant
  Graft loss is defined by initial engraftment (assessed by neutrophil recovery and donor chimerism) with the subsequent loss of donor myeloid chimerism (regardless whether persistent neutropenia develops).
Number of Participants Experiencing Cytomegalovirus (CMV) Viremia | Up to Day 180
  Cytomegalovirus (CMV) viremia is defined as positive blood antigen or polymerase chain reaction (PCR) test.
Number of Participants Experiencing CMV Invasive Disease | 1 year post-transplant
  CMV invasive disease is defined in accordance with the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures.
Number of Participants Experiencing Post-transplant Lymphoproliferative Disorder (PTLD) | 1 year post-transplant
  Post-transplant lymphoproliferative disorder (PTLD) is defined in accordance with the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures and the World Health Organization's Classification of Tumours of Haematopoietic and Lymphoid Tissues.
Number of Participants Experiencing Other Infections | 1 year post-transplant
  Infections other than CMV viremia, CMV invasive disease, and PTLD is defined in accordance with the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures.
Number of Participants Experiencing Immune Reconstitution | 1 year post-transplant
  Immune reconstitution is assessed by the day 100 cluster of differentiation 4 (CD4+) T cell count and by the reaccumulation of natural killer (NK) cells, B cells, total T cells, and cluster of differentiation 8 (CD8+) T cells as assessed by multicolor flow cytometry.
Number of Participants Experiencing Acute Graft Versus Host Disease (GVHD) | Up to 1 year post-transplant
  Early onset (before day 100) and late onset (after day 100) acute GVHD is assessed according to the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures using the NIH consensus criteria.
Number of Participants Experiencing Chronic GVHD | 2 years post-transplant
  Chronic GVHD, including overlap syndrome, is assessed according to the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures using the NIH consensus criteria.
Immune Suppression-Free Survival Rate | 1 year post-transplant
  Participant survival while off of immunosuppressive agents.
Immune Suppression-Free and Disease-Free Survival Rate | 1 year post-transplant
  Participant disease-free survival while off of immunosuppressive agents.
Disease-free Survival Rate | 1 year post-transplant
  Disease-free survival is defined as survival without recurrence of underlying disease.
Overall Survival Rate | 1 year post-transplant
  Overall-survival is defined as survival with or without relapse of underlying disease

CONTACTS AND LOCATIONS:
Overall Officials: John T Horan, MD, Principal Investigator — Children's Healthcare of Atlanta/Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States